CLINICAL TRIAL: NCT03121651
Title: Medication Management Among Individuals With Neurodevelopmental Disabilities
Acronym: M-MIND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Karen Farris, PhD., Charles R. Walgreen III Professor of Pharmacy Administration, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: HUM00107874 and HUM00139267; 90RE5012 (Other Grant/Funding Number: NIDILRR)
Record Dates: First submitted 2017-04-07; First posted 2017-04-20 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Spina Bifida; Cerebral Palsy
Keywords: Mobile technology; Reinforcement-learning; Medication management
MeSH Terms: conditions — Spinal Dysraphism; Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Unblinded pilot study with 1 intervention arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RL-adaptive application (Experimental): Dyad is comprised of individual with disability (spina bifida or cerebral palsy) and the respective parent/legal guardian (also referred to as caregivers).
  Young adult will use the RL-adaptive support application that the investigators are developing to help manage medications.
  Interventions: Device: RL-adaptive application

INTERVENTIONS:
Device: RL-adaptive application — Up to 6 dyads of individuals with disabilities and their caregivers will be recruited to collaborate in defining the features and content of the RL-adaptive support. The steps in developing the RL-adaptive support include having the dyads use for approximately 6 weeks each:
  1. young adult uses an electronic medication pillbox that sends its pillbox openings within one hour of opening to the research team,
  2. young adult uses the electronic medication pillbox + both use a commercially available medication reminder app + caregiver uses a pillbox opening notification app, and
  3. young adult uses the electronic medication pillbox + the RL-adaptive support including push notifications in the form of text messages + caregiver uses the pillbox opening notification app.
  The goal is to reduce the number of caregiver prompts necessary for the medication pillbox to be opened.

SUMMARY:
This is a pilot study to develop a reinforcement learning (RL)-adaptive visual and interactive support application (hereafter RL-adaptive support) to help young adults with spina bifida or cerebral palsy become more independent with medication management. Individuals with disabilities who are empowered to manage several aspects of their lives can ultimately be better integrated into and contribute more to society.

DETAILED DESCRIPTION:
In this study, an application will be iteratively developed and tested using RL-adaptive support for young adults with disabilities, with the goal to promote the transition to independent self-medication administration among young adults with cerebral palsy and spina bifida.

Stochastic mathematical models of how individuals with varying levels of executive function and psychomotor skills will respond to the interventions (i.e. the different types and formats of messages) of the RL-adaptive support will be developed.

Up to 6 dyads of individuals with disabilities and their caregivers were intended to be recruited to collaborate in defining the features and content of the RL-adaptive support. The investigators recruited 3 dyads.

The steps in developing the RL-adaptive support include having the dyads use for approximately 6 weeks each:

1. young adult uses an electronic medication pillbox that sends its pillbox openings within one hour of opening to the research team,
2. young adult uses the electronic medication pillbox + both use a commercially available medication reminder app + caregiver uses a pillbox opening notification app, and
3. young adult uses the electronic medication pillbox + the RL-adaptive support including push notifications in the form of text messages + caregiver uses the pillbox opening notification app

The goal was to reduce the number of caregiver prompts necessary for the medication pillbox to be opened. Using these data, the number and type of prompts necessary for the caregiver to open the electronic pillbox can be determined. In case the young adult does not open the electronic pillbox within two hours, the caregiver will be notified so that pills are not missed. In each step, the useful features of the system will be determined via qualitative and quantitative feedback with specific suggestions about how to improve this supportive system.

ELIGIBILITY:
Inclusion Criteria:

For young adult:

* Diagnosed with cerebral palsy or spina bifida and previously enrolled in HUM00081812
* Age 18-26 years-old
* Having mild-moderate cognition based on consultation with the investigators and the results of the following tests: iBRIEF Metacognition index T-Score, CVLT List A Free Recall T Score, ReyO Organization T-Score, PPVT Scaled Score, Tower Scaled Score, TRAQ question 4: Do participants take medications correctly and on their own?
* Having adequate physical dexterity (to be able to open a pill box and use an iPad/tablet)
* Taking two or more routine oral medicines in pill formulation
* Being able to take capsules or tablets
* Still living at home with their parent/legal guardian
* Have Wi-Fi/Internet access at home

For parent/caregiver:

* Being the parent/legal guardian of a person with aforementioned disability
* Owning a cell phone
* Have Wi-Fi/Internet access at home

Exclusion Criteria:

• Those who do not fulfill the inclusion criteria will be excluded from the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Prefer to continue to use RL-adaptive support after study is over | at least 18 weeks after beginning study
  Qualitative feedback

SECONDARY OUTCOMES:
Usefulness of the aspects of the RL-adaptive support | End of each phase, which lasts approximately 6 weeks
  Qualitative feedback
Most and least helpful aspects of RL-adaptive support application | End of each phase, which lasts approximately 6 weeks
  Qualitative feedback
Ease of use of RL-adaptive support application | End of each phase, which lasts approximately 6 weeks
  Qualitative feedback

CONTACTS AND LOCATIONS:
Overall Officials: Karen B Farris, PhD, Principal Investigator — Professor and Chair, Department of Clinical Pharmacy, University of Michigan College of Pharmacy
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD